CLINICAL TRIAL: NCT02931812
Title: Feeding Behavior and Taste Sensitivity Before and After Liver or Renal Transplantation
Acronym: GREFFE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Burgundy (Other)
Responsible Party: Principal Investigator, Laurent BRONDEL, Professor, University of Burgundy
Other Study IDs: 2014-A00254-43
Record Dates: First submitted 2016-10-03; First posted 2016-10-13 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Cirrhosis; Food Preferences; Taste Disorders; Protein-Energy Malnutrition; Chronic Renal Failure
Keywords: cirrhosis; reward system; taste sensitivity; chronic renal failure
MeSH Terms: conditions — Fibrosis; Food Preferences; Taste Disorders; Protein-Energy Malnutrition; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for hormones measurments (leptine, ghrelin, insulin) and plasmatic amino-acids
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Cirrhotic subjects: 15 cirrhotic patients in end-stage in waiting a graft
- Chronic kidney disease subjects: 15 chronic kidney disease patients in end-stage in waiting a graft
- Healthy subjects: 30 healthy subjects to compare

SUMMARY:
This study evaluates the influence of the taste sensitivity, of food preferences and of the reward system on the energetic balance before and after liver transplantation in cirrhotic patients and after kidney transplantation in renal failure patients

DETAILED DESCRIPTION:
Background and Aims: Protein-energy malnutrition is associated to cirrhosis with a high prevalence and greatly increases the morbidity and mortality of the disease. Malnutrition results of numerous causes including intestinal malabsorption, increased energy resting expenditure, metabolism disturbances, impaired sensory taste and changes in food preferences which might participate to a reduction in food intake. The aim of this study was to determine the relationships that may exist between taste sensitivity and food preferences on the one hand, eating habits, nutritional status, energy balance and biological parameters including amino acids on the other hand in patients with end-stage cirrhosis and in patients with renal failure.

Fifteen end-stage cirrhotic patients and 15 renal failure patients will be included and matched with 30 healthy subjects. The following parameters will be evaluated during a morning testing session: gustatory sensitivity using a triangular detection threshold method for sweet, salty and umami solutions; preferences for fat- and carbohydrate-rich foods using the PrefQuest score; liking for six foods (protein-, carbohydrate- and fat-rich foods) and wanting for 18 foods (photographs); hunger sensation; energy intake (24 h ingested food); body composition (BMI and impedancemetry); resting energy expenditure (indirect calorimetry) and physical activity (questionnaire). Several plasmatic parameters (amino-acids, leptin, ghrelin, lipid profile) will be also determined.

ELIGIBILITY:
Inclusion Criteria:

* written consent
* patients in waiting renal transplant
* patients in waiting liver transplant

Exclusion Criteria:

* chronic infection
* acute infection
* cancer
* antibiotic treatments
* alcool abuse
* pregnant woman
* specific or restrictive diet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 15 patients waiting for renal transplantation
  * 15 patients waiting for liver transplantation
  * 30 healthy subjects matched for gender, age and body mass index
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-05; Primary Completion 2020-05 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure | two years
  evice: indirect calorimetry (sensormedics)
body composition | 2 years
  Device: Multifrequency bio-impedancemetry (aminostats)
amino acids profil in plasma | 2 years
  Biological measurments
Food preferences | 2 years
  Device: Treshold taste detection

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Taste and Feeding Behaviour, Dijon, Burgundy, France

IPD SHARING:
Plan to Share IPD: No